CLINICAL TRIAL: NCT07324876
Title: A Multicenter Real-World Study on TKI Therapy After Progression on First-Line TKI/IO Therapy or TKI/IO Therapy After Progression on First-Line TKI in Chinese Patients With Metastatic Renal Cell Carcinoma (mRCC)
Status: Not yet recruiting | Type: Observational
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: E20250713
Record Dates: First submitted 2025-12-23; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: RCC
Keywords: tyrosine kinase inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- the TKI/IO-TKI sequential treatment group
- the TKI-TKI/IO sequential treatment group

SUMMARY:
TKI monotherapy or TKI/IO combination therapy is the standard first-line treatment for low- and intermediate-risk advanced renal cell carcinoma (RCC). In clinical practice, after the failure of first-line therapy, sequential treatment is often selected based on the initial regimen, with options including TKI/IO therapy or TKI therapy. In the real-world setting of low- and intermediate-risk advanced RCC in China, which sequential treatment strategy-TKI/IO-TKI or TKI-TKI/IO-provides greater survival benefits for patients? This study aims to compare the efficacy, safety, and cost-effectiveness of TKI/IO-TKI sequential therapy versus TKI-TKI/IO sequential therapy in real-world low- and intermediate-risk mRCC patients. The objective is to accurately identify the optimal patient subgroups for each treatment strategy, optimize treatment plans, improve patient quality of life, reduce healthcare costs, provide guidance and reference for the clinical management of low- and intermediate-risk mRCC patients, and contribute to the refinement and updating of related Chinese treatment guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with histologically confirmed unresectable metastatic renal cell carcinoma (mRCC) will be included in the study. Previous nephrectomy or metastasectomy is allowed, but no prior systemic anticancer therapy targeting RCC is permitted.
2. Classified as low- or intermediate-risk according to the International Metastatic Renal Cell Carcinoma Database Consortium (IMDC) criteria.
3. Male or female subjects aged 18 years or older at the time of signing the informed consent form.
4. Defined as Chinese ethnicity, with both biological parents and all four biological grandparents being of Chinese descent.
5. Patients who progressed or were intolerant to first-line TKI therapy (including sunitinib, pazopanib, cabozantinib, sorafenib, axitinib, lenvatinib, etc.) and subsequently received TKI/IO therapy (including axitinib/ lenvatinib/ cabozantinib combined with toripalimab/ tislelizumab/ pembrolizumab/ sintilimab/ nivolumab, etc.).
6. Patients who progressed or were intolerant to first-line TKI/IO therapy (including axitinib/ lenvatinib/ cabozantinib combined with toripalimab/ tislelizumab/ pembrolizumab/ sintilimab/ nivolumab, etc.) and subsequently received TKI therapy (including sunitinib, pazopanib, cabozantinib, sorafenib, axitinib, lenvatinib, etc.).
7. Karnofsky Performance Status (KPS) ≥ 70% within 10 days prior to the first dose of treatment.
8. Adequate organ function as evidenced by laboratory values: ANC ≥ 1500/μL; platelets ≥ 100,000/μL; hemoglobin ≥ 10.0 g/dL or ≥ 6.2 mmol/L; CrCl ≥ 30 mL/min; AST and ALT ≤ 2.5 × ULN; total bilirubin ≤ 1.5 × ULN; and INR or PT ≤ 1.5 × ULN.

Exclusion Criteria:

1. Requiring intermittent oxygen supplementation at rest, or long-term oxygen therapy.
2. Clinically significant cardiovascular disease within 6 months prior to the first dose of study intervention.
3. Severe active, non-healing wound, ulcer, or fracture.
4. Use of colony-stimulating factors (e.g., G-CSF, GM-CSF), recombinant erythropoietin (EPO), or blood transfusion within 28 days prior to the first dose of study intervention.
5. Inability to swallow oral medications or a history of, or current evidence of, gastrointestinal diseases (e.g., inflammatory bowel disease, Crohn's disease, ulcerative colitis) or impaired liver function, or other conditions that, in the investigator's opinion, may significantly alter the absorption or metabolism of oral study interventions.
6. Severe hypersensitivity reactions to TKI drugs, IO drugs, and/or any excipients.
7. Diagnosis of immunodeficiency or use of long-term systemic corticosteroids (daily dose exceeding 10 mg prednisone or equivalent) or any form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
8. Diagnosis of another malignancy (excluding RCC treated by nephrectomy and/or metastasectomy) that is currently progressing or required active treatment in the past 3 years. Note: Subjects with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (excluding bladder carcinoma in situ) who have undergone potentially curative treatment are eligible.
9. Active autoimmune disease requiring systemic treatment (i.e., use of disease-modifying agents, corticosteroids, or immunosuppressive drugs) within the past 2 years. Replacement therapy (e.g., thyroxine, insulin, or physiological corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered systemic treatment and is allowed.
10. History of or current (non-infectious) pneumonitis/interstitial lung disease requiring steroid treatment, or current pneumonitis/interstitial lung disease.
11. Active infection requiring systemic treatment.
12. Known history of HIV infection, hepatitis B (defined as HBsAg reactive), or active hepatitis C virus (defined as detectable HCV RNA [qualitative]). Note: Testing for HIV, HBV, or HCV is not required unless mandated by local health regulations.
13. Any prior or current condition, treatment, laboratory abnormality, or other circumstance that may interfere with the study results, affect the subject's ability to complete the study, or, in the investigator's opinion, make the subject unsuitable for participation or unlikely to benefit from the study.
14. Known psychiatric or substance abuse disorders that would interfere with the subject's ability to comply with study requirements
15. History of prior allogeneic tissue/solid organ transplantation.
16. If the subject is a non-pregnant and non-lactating female, the subject must agree to use highly effective (failure rate <1% per year) and low-dependency contraceptive methods during treatment.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Renal cell carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 860 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS2 | 1year
  defined as the time from the initiation of first-line treatment to disease progression on second-line therapy or death from any cause in a real-world setting

SECONDARY OUTCOMES:
1L-rwPFS | 1year
  Evaluate the real-world progression-free survival of first-line therapy (1L-rwPFS) for both cohorts
2L-rwPFS | 1year
  Evaluate the real-world progression-free survival of second-line therapy (2L-rwPFS) for both cohorts
OS | 1year
  the overall survival
ORR | 1year
  Assess the objective response rate (ORR) of primary and metastatic lesions based on RECIST 1.1 criteria for both cohorts
saftey | 1year
  Evaluate the safety profiles of the treatments in both cohorts

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: Undecided